CLINICAL TRIAL: NCT03610945
Title: A Non-Randomized, Open-Label, Two-Part, Drug-Drug Interaction Study to Evaluate the Effects of Fluconazole and Quinidine on the Pharmacokinetics and Safety of EDP-305 in Healthy Volunteers
Brief Title: Drug-drug Interaction Study Between EDP-305, Fluconazole and Quinidine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 305-007
Record Dates: First submitted 2018-07-12; First posted 2018-08-01 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: drug-drug interaction
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fluconazole; Quinidine; EDP-305

STUDY DESIGN:
Intervention Model Description: 2-Part Single Group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDP-305 and fluconazole interaction (Part 1) (Experimental)
  Interventions: Drug: Fluconazole; Drug: EDP-305
- EDP-305 and quinidine interaction (Part 2) (Experimental)
  Interventions: Drug: Quinidine; Drug: EDP-305

INTERVENTIONS:
Drug: Fluconazole — Subjects will receive fluconazole once daily from Day 5 to Day 18
  Arms: EDP-305 and fluconazole interaction (Part 1)
Drug: Quinidine — Subjects will receive quinidine twice daily from Day 5 to Day 12
  Arms: EDP-305 and quinidine interaction (Part 2)
Drug: EDP-305 — Subjects will receive a single dose of EDP-305 on Day 1 and Day 14
  Arms: EDP-305 and fluconazole interaction (Part 1)
Drug: EDP-305 — Subjects will receive a single dose of EDP-305 on Day 1 and Day 8
  Arms: EDP-305 and quinidine interaction (Part 2)

SUMMARY:
This is a non-randomized, 2-part, open-label, drug-drug interaction (DDI) study to evaluate the effect of concomitant administration of fluconazole or quinidine on the pharmacokinetics and safety of EDP-305 in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Female subjects must be of non-childbearing potential.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.
* Clinically significant electrocardiogram abnormalities or QTcF greater than 450 ms for males and 470 ms for females at either Screening or Day -1 (Part 2 only), or any prior history of QT abnormality.
* For Part 2 subjects, the following cardiovascular abnormalities

  * QRS duration >110 ms
  * Incomplete right bundle branch block or any complete bundle branch block
  * Heart rate <40 or >90 beats per minute (per vital sign capture while rested)
  * History of unexplained syncope, structural heart disease, or clinically significant arrhythmias
  * Personal or family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome
  * PR interval >220 ms or any 2nd or 3rd degree AV block
  * Ventricular pre-excitation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-305 with and without coadministration with fluconazole | Up to 19 days
AUC of EDP-305 with and without coadministration with fluconazole | Up to 19 days
Cmax of EDP-305 with and without coadministration with quinidine | Up to 13 days
AUC of EDP-305 with and without coadministration with quinidine | Up to 13 days

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No